CLINICAL TRIAL: NCT02527616
Title: A Randomised, Crossover Investigation to Evaluate and Compare the Effectiveness, Safety and Feasibility of a Novel Dedicated Over-The-Wire FFR Infusion Microcatheter (HYPEREM™IC) for Measuring Fractional Flow Reserve (FFR) Using Intra-coronary Non-weight Adjusted Adenosine Infusion With the Standard Intra-venous Administration of Adenosine, in Subjects With Intermediate Coronary Artery Stenosis.
Brief Title: An Investigation to Evaluate an Over-The-Wire FFR Infusion Microcatheter (HYPEREM™IC) for Measuring Fractional Flow Reserve (FFR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diasolve Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: DIAS-001-FFR
Record Dates: First submitted 2015-08-05; First posted 2015-08-19 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV followed by IC (investigation) (Experimental): The patient undergoes the FFR measurement with the standard measurement first followed by FFR measurement using the FFR Infusion Microcatheter
  Interventions: Device: FFR Infusion Microcatheter and standard intra-venous (IV) infusion
- IC (investigation) followed by IV (Experimental): The patient undergoes the FFR measurement using the FFR Infusion Microcatheter measurement first followed by measurement via the standard measurement
  Interventions: Device: FFR Infusion Microcatheter and standard intra-venous (IV) infusion

INTERVENTIONS:
Device: FFR Infusion Microcatheter and standard intra-venous (IV) infusion — Cross-over design where FFR is measured twice in the same lesion using standard standard intra-venous (IV) infusion and new method
  Other Names: HYPEREM™IC; REF: 143836-01 GTIN: 5060420320008.; HYPERAEM

SUMMARY:
This is a single-blinded, randomised, crossover investigation comparing the investigational device using intra-coronary (IC) Adenosine infusion to the standard intra-venous (IV) infusion method used for obtaining FFR measurements. All subjects requiring on a clinical basis a pressure wire assessment of intermediate coronary artery stenosis(es) will be eligible to take part in the investigation.

DETAILED DESCRIPTION:
Coronary artery disease is the most common type of heart disease that affects millions of people worldwide. It is caused by a narrowing or blocking of the arteries (known as stenosis) due to plaque, which restricts blood flow and reduces the amount of oxygen to the heart.

Over the past decade, fractional flow reserve (FFR) measurement has been increasingly used in cardiac catheterization laboratories, providing a straightforward and readily available quantitative assessment of the functional severity of a coronary artery stenosis, as the ability of the cardiologist to discriminate between stenoses that can cause ischemia and those that are physiologically insignificant on the basis of coronary angiography alone is limited.

Measuring FFR determines the ratio between the maximum achievable blood flow in a diseased or narrowed coronary artery and the maximum blood flow in a normal coronary artery. This ratio represents the potential decrease in coronary flow distal to the coronary stenosis.

FFR is easily measured during routine coronary angiography by using a pressure wire to calculate the ratio between the coronary pressure distal to a stenosis or a diseased segment and the aortic pressure under conditions of maximum myocardial hyperemia. An FFR of 1.0 is widely accepted as normal. An FFR lower than 0.80 is generally considered to be associated with coronary ischemia and widely accepted in favour of revascularization over conservative management.

The current standard methods of measuring FFR is to insert a pressure wire into the coronary artery while the hyperaemic agent, normally adenosine, is delivered by continuous intravenous infusion via a central femoral vein, a large ante-cubital peripheral cannula or intra-coronary bolus injection.

The investigational device in this clinical investigation is an FFR catheter being developed by Diasolve Limited; a UK based medical device development company. The FFR catheter is a combined pressure wire and hyperaemic agent delivery catheter, which allows simultaneous delivery of a pressure wire and administration of the hyperaemic agent directly into the coronary ostium or most proximal section of the coronary artery, when performing a FFR measurement using currently available pressure wire systems such as Pressure Wire Certus or Prestige from St Jude Medical.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give written informed consent prior to investigation participation.
2. Has given consent to undergo hospital's diagnostic or interventional coronary procedure.
3. Male and female subjects aged 18 and over.
4. Ability to communicate well with the investigator and to comply with the requirements of the clinical investigation.

Prior to randomisation:

1. Coronary angiogram demonstrates at least one coronary stenosis of intermediate severity (40-70%), in a non-infarct related artery, which requires FFR measurement for physiological assessment.

-

Exclusion Criteria:

1. Known sensitivity to adenosine or any of its excipients
2. Technically inaccessible stenosis(es)
3. Acute ST segment elevation myocardial infarction (STEMI)
4. Haemodynamically unstable
5. Presence of any clinically significant medical condition as determined by the investigator
6. Participation in another clinical investigation within the three months prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with comparable FFR ratio recordings | Intraoperative
  The FFR ratio should remain constant when measured by the standard method and the investigational device.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Intraoperative
  Participants should not experience any additional adverse events during FFR ratio measurement using the investigational device than they do using the standard method.
Dose of adenosine administered. | Intraoperative
  Maximum hyperaemia may be achieved with a reduced dose of adenosine using the FFR Catheter.
Time to onset of maximum hyperaemia. | Intraoperative
  Maximum hyperaemia may be achieved faster using the FFR Catheter

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elghamaz, MB BCh, MRCP, Principal Investigator — London North West Healthcare NHS Trust; Paul Wenberger, Study Chair — Diasolve Ltd
Locations (1):
- Northwick Park Hospital, Harrow, Middx, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual data will not be shared